CLINICAL TRIAL: NCT06924593
Title: Study on the Safety and Efficacy of the Trans-Carotid Artery Occlusion Shunt System for Carotid Artery Revascularization During Endovascular Treatment
Brief Title: Study on the Trans-Carotid Artery Occlusion Shunt System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Wecan Medical Technology Co.,Ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: WKP002CT(CN)-01
Record Dates: First submitted 2025-04-06; First posted 2025-04-11 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-04

CONDITIONS: Revascularization; Carotid Artery Stenosis; Carotid Artery Diseases
MeSH Terms: conditions — Carotid Stenosis; Carotid Artery Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trans-Carotid Artery Occlusion Shunt System (Experimental): Device systems for Carotid Artery Revascularization during Endovascular Treatment
  Interventions: Device: Trans-Carotid Artery Occlusion Shunt System

INTERVENTIONS:
Device: Trans-Carotid Artery Occlusion Shunt System — To evaluate the Safety and Efficacy of the Trans-Carotid Artery Occlusion Shunt System for Carotid Artery Revascularization during Endovascular Treatment

SUMMARY:
The objective of the study is to evaluate the Safety and Efficacy of the Trans-Carotid Artery Occlusion Shunt System for Carotid Artery Revascularization during Endovascular Treatment

DETAILED DESCRIPTION:
The physician shall strictly follow the clinical study protocol and shall not deviate from or substantially change the protocol. However, in case of emergency such as immediate risk to the subjects, which needs tobe eliminated immediately, it may be reported in written form afterwards. During the course of the study,documents such as amendments to the clinical study protocol and informed consent, requests for deviation,and resumption of the suspended clinical study shall be subject to the written approval of the Ethics Committee

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* For patients diagnosed with carotid artery stenosis and planned to undergo transcarotid artery endovascular revascularization, one of the following conditions must be met:

  1. Symptomatic carotid artery stenosis: The degree of stenosis is determined by non-invasive imaging or angiography to be > 50%, and the patient has a history of stroke (mild or non-disabling), transient ischemic attack (TIA), and/or amaurosis fugax within 180 days before the operation.
  2. Asymptomatic carotid artery stenosis: The degree of stenosis is determined by non-invasive imaging or angiography to be > 70%, and the patient has not experienced any neurological symptoms within 180 days before the operation.
* The modified Rankin Scale (mRs) score ≤ 2 before enrollment.
* The patient must meet at least one of the following important anatomical or comorbid high-risk conditions in order to be included in the study:

Anatomical high-risk:

A. Contralateral carotid artery occlusion; B. Presence of tandem stenosis in the internal carotid artery with a stenosis degree > 70%; C. Carotid artery stenosis above the C2 vertebral body; D. Restenosis after previous ipsilateral carotid endarterectomy; E. Bilateral carotid artery stenosis requiring treatment (treatment of the contralateral vessel should be carried out at least 30 days after the operation); F. "Difficult neck" suitable for the transcarotid approach as evaluated by the researcher, including but not limited to: history of previous neck radiotherapy, history of previous radical neck lymph node dissection, neck stoma or limited cervical spine mobility.

Comorbid high-risk:

G. The patient's age is ≥ 70 years old; H. The patient has coronary artery disease involving > 2 vessels and has a history of angina pectoris of any severity; I. The patient has a history of angina pectoris, with Canadian Cardiovascular Society (CCS) angina class 3 or 4, or unstable angina pectoris (defined as resting angina pectoris accompanied by electrocardiogram changes); J. The patient has congestive heart failure (CHF) - New York Heart Association (NYHA) functional class 3 or 4; K. The patient is known to have severe left ventricular dysfunction with a left ventricular ejection fraction (LVEF) < 30%; L. The patient has experienced a myocardial infarction within 72 hours to 6 weeks before the operation; M. The patient has severe pulmonary disease (chronic obstructive pulmonary disease, COPD), with a forced expiratory volume in one second (FEV1) < 50% (predicted value), or has been receiving long-term oxygen therapy, or has an arterial partial pressure of oxygen (PO2) ≤ 60 mmHg (room air) at rest; N. The patient has permanent contralateral cranial nerve injury; O. The patient has chronic renal insufficiency (serum creatinine > 2.5 mg/dL).

* The diameter of the common carotid artery on the target lesion side is > 6 mm;
* The patient is able to understand the purpose of the trial, voluntarily participates in this study, signs the informed consent form, and is willing to complete the follow-up according to the requirements of the protocol.

Exclusion Criteria:

* Anatomical exclusion criteria:

There are extensive atherosclerotic plaques in the proximal part of the common carotid artery on the target lesion side, making the safe operation of the surgery difficult; There are lesions in the access area of the common carotid artery on the target lesion side and its proximal part towards the heart; The distance from the superior border of the clavicle on the target lesion side to the bifurcation of the common carotid artery is less than 5 cm; A stent or graft has been implanted in the carotid artery on the target lesion side; There are acute or subacute thrombosis, arteriovenous malformations at the target lesion or adjacent areas; Severe calcification or tortuosity at the target lesion site makes it difficult to deliver the instruments to the designated location; The target carotid artery is completely occluded;

* Known to have uncontrollable hypertension (systolic blood pressure continuously ≥ 180 mmHg or diastolic blood pressure continuously ≥ 110 mmHg);
* Combined with symptomatic severe stenosis of other blood vessels (including intracranial and extracranial vessels);
* The patient has experienced an ischemic stroke within 3 months, and the stroke affects the evaluation of the endpoints;
* There has been spontaneous intracranial hemorrhage within 12 months;
* Carotid artery stenosis not caused by atherosclerosis (such as dissection, fibromuscular dysplasia, etc.);
* There are other heart diseases that may lead to embolism: such as left ventricular aneurysm, intracardiac filling defect, cardiomyopathy, artificial aortic valve or artificial mitral valve, calcific aortic stenosis, endocarditis, mitral stenosis, atrial septal defect, atrial septal aneurysm or left atrial myxoma, etc.;
* Severe dementia or other nervous system diseases that may interfere with the evaluation of neurological function;
* Advanced heart failure;
* Chronic atrial fibrillation; Paroxysmal atrial fibrillation with an episode within 6 months or paroxysmal atrial fibrillation requiring long-term anticoagulant therapy;
* Myocardial infarction occurred within 72 hours before the operation;
* Coronary artery bypass grafting (CABG), endovascular stent surgery, cardiac valve surgery or vascular surgical procedures have been or will be performed within 30 days before and after the operation;
* There is an active bleeding tendency or severe coagulation dysfunction; There has been gastrointestinal bleeding within 30 days before the operation, which will affect antiplatelet therapy;
* Hemoglobin (Hgb) < 8 gm/dL, platelet count < 90×10^9/L or a history of heparin-induced thrombocytopenia;
* Patients with abnormal liver and kidney function before the operation [Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) exceeding 5 times the upper limit of the normal value; Serum creatinine (Cr) > 3.0mg/dL (265.2μmol/L) or end-stage renal disease receiving hemodialysis];
* Patients known to be allergic to contrast agents, stent and delivery device materials (referring to nitinol, PTFE, nylon polymer materials); Patients known to have contraindications to anticoagulant and antiplatelet drugs;
* Intracranial tumors or other malignant tumors;
* Life expectancy is less than 1 year;
* Women who plan to become pregnant, are pregnant or are breastfeeding;
* Patients who are participating in other clinical trials at the same time and have not withdrawn from the trials;
* Patients who are judged by the researcher as not suitable for participating in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The composite incidence rate of death, stroke, and myocardial infarction within 30 days after the operation. | 30 days after the operation
  The composite incidence rate of death, stroke, and myocardial infarction.

SECONDARY OUTCOMES:
Immediate technical success rate | Immediate technical success rate
  Immediate technical success is defined as complete occlusion of the proximal common carotid artery, effectively establishing a blood flow reversal circulation pathway, and successfully withdrawing the device.
Surgical success rate | 30 days after the operation
  Surgical success is defined as technical success without major adverse events (MAE is defined as death, stroke, or myocardial infarction).
Incidence rate of stroke within 30 days after the operation | 30 days after the operation
  The researcher will confirm whether the subject has suffered a stroke.
Incidence rate of cranial nerve injury within 30 days after the operation | 30 days after the operation
  The researcher will confirm whether the subject has suffered a cranial nerve injury.
Incidence rate of myocardial infarction within 30 days after the operation | 30 days after the operation
  The researcher will confirm whether the subject has suffered a myocardial infarction.
All-cause mortality rate within 30 days after the operation | 30 days after the operation
  All-cause mortality refers to deaths from any cause that occur within the follow-up time points.
Incidence rate of access complications within 30 days after the operation | 30 days after the operation
  Access complications refer to various adverse situations or complications that occur during or after the establishment of vascular accesses.
Incidence rate of ipsilateral stroke within 30 days after the operation | 30 days after the operation
  The researcher will confirm whether the subject has suffered a ipsilateral stroke.
Device-related adverse events | Before discharge (up to 14 days), 30 days after the operation
  Adverse events refer to adverse medical events that occur during the process of a clinical trial, regardless of whether they are related to the medical device used in the trial. However, normal postoperative stress responses should be distinguished, such as fever, discomfort in the chest and back, etc. If, upon the judgment of the researcher, it is determined to be a normal postoperative stress response, there is no need to record it as an adverse event of the medical device. Adverse events related to the medical device refer to situations that are determined by the researcher to be definitely related, possibly related, or undeterminable in relation to the medical device used in the trial.
Incidence rate of serious adverse events | Before discharge (up to 14 days), 30 days after the operation
  Serious adverse events refer to events that occur during the clinical trial process and lead to death or a serious deterioration of health status, including fatal diseases or injuries, permanent defects in body structure or body function, the need for hospitalization or an extended hospital stay, the need to take medical measures to avoid permanent defects in body structure or body function, and events that lead to fetal distress, fetal death, or congenital abnormalities and congenital defects.

CONTACTS AND LOCATIONS:
Overall Officials: zhong chen, Professor, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No